CLINICAL TRIAL: NCT05198765
Title: Reducing Clinical Inertia in Obesity Management of Diabetes Patients in Primary Care: Cluster-Randomized Trial
Brief Title: Weight Loss Clinical Decision Support
Acronym: BMI-CDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-107; 1R01DK128281-01 (NIH)
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Clinical Decision Support; Shared Decision Making; Diabetes; Metabolic Bariatric Surgery; Obesity Management; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI-CDS (Experimental): Clinicians and their patients assigned to intervention clinics will receive shared decision support tools for weight loss management.
  Interventions: Behavioral: BMI-CDS
- Usual Care (No Intervention): Clinicians and their patients assigned to control clinics will engage in the usual standard of care.

INTERVENTIONS:
Behavioral: BMI-CDS — The BMI-CDS is a sophisticated point of care shared decision support tool for patients with type 2 diabetes and high BMI. The intervention is built on existing point of care clinical decision support system that algorithmically identifies study-eligible patients and deploys patient-specific CDS output at an index visit and updated CDS all subsequent primary care office, video, and phone encounters.
  Other Names: Weight Loss Wizard; BMI Wizard
  Arms: BMI-CDS

SUMMARY:
Despite steady increases in obesity prevalence, the more than 12 million obese U.S. adults with type 2 diabetes (T2DM) and severe obesity encounter a number of barriers to adopting effective surgical and pharmaceutical treatments, including: (a) both patients and primary care clinicians frequently underestimate the effectiveness and potential benefits of obesity treatments; and (b) both patients and clinicians typically lack access to evidence-based estimates of the patient-specific potential benefits and risks of appropriate obesity treatment options. This project addresses these important obstacles to evidence-based obesity care by providing accurate, patient-specific estimates of benefits and risks of various obesity treatment options to inform shared decision making about obesity treatment.

In this project the study team will implement a scalable, web-based point-of-care decision-support intervention in primary care that provides patient-specific estimates of obesity treatment benefits and risks in a randomized trial in 40 primary care clinics with 15,810 eligible patients, and assess intervention impact on (i) appropriate active management of obesity in eligible patients, (ii) weight trajectories, and (iii) patient and clinician satisfaction with the decision support intervention.

DETAILED DESCRIPTION:
Obesity has been steadily increasing in prevalence and now affects more than 4 in 10 U.S. adults, leading to many adverse health outcomes including myocardial infarction, stroke, type 2 diabetes (T2DM), hypertension, sleep apnea, arthritis, and others. Effective surgical, pharmaceutical, and behavioral treatments for obesity are available, and the evidence to support the broad use of these treatments for obesity is very well established. However, active management of obesity defined as prescribing or referring adults with obesity for lifestyle, pharmaceutical, or surgical treatment of obesity, is greatly underused. Major underlying reasons for underutilization of effective obesity treatments include: (a) both patients and primary care clinicians (PCCs) frequently underestimate the effectiveness and potential benefits of obesity treatments; and (b) both patients and clinicians typically lack access to evidence-based, patient-specific estimates of the potential benefits and risks of appropriate patient-specific obesity treatment options.

To address this problem, the study team will integrate externally validated prediction equations that estimate benefits and risk of various obesity treatment options in adults with T2DM into a widely-used and successful clinical decision support system in order to deliver appropriate patient-specific obesity treatment suggestions at the point of care. The team will implement a scalable, web-based point-of-care decision-support intervention in a randomized trial in 40 primary care clinics with 15,810 eligible patients, and assess intervention impact on the following primary outcomes: (a) appropriate referral of eligible patients for evaluation for metabolic bariatric surgery (MBS); (b) appropriate initiation of FDA-approved medications for weight loss; (c) weight trajectories; and (d) patient-reported conversations with their PCC about weight loss and intentions to engage in weight loss. In addition, the study team collect and analyze clinician-reported and patient-reported data to identify factors that may impede or facilitate broad dissemination of this intervention strategy to other care delivery settings.

This innovative project will (a) provide state-of-the-art scientific evidence on obesity treatment to large numbers of obese American adults with T2DM and their PCCs at the point of care; (b) help PCCs identify appropriate patient-specific obesity treatment options; (c) implement in primary care a web-based electronic health record (EHR)-linked obesity treatment clinical decision support model that uses state-of-the-art Health Information Technology (HIT) standards, is broadly scalable, easy to update as evidence changes, and optimized for clear communication of information to patients and PCCs; and (d) improve the clinical return on ongoing massive private and public investments in outpatient health information systems.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18-75 years at index clinical encounter)
* Existing diagnosis of T2DM
* BMI ≥35 kg/m2 at index clinical encounter
* Have an index clinical encounter with a PCC (family practice or general internal medicine physician, nurse practitioner, or physician assistant) at a randomized study clinic during a 12-month accrual period

Exclusion Criteria:

* Prior MBS
* Patients diagnosed with cancer (except non-melanoma skin cancer), dementia, and/or cirrhosis.
* Pregnant or breastfeeding.
* In long-term care, palliative care, or hospice care.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10120 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients referred to an MBS program | Within 18 months of index visit date
  Proportion of study-eligible patients with estimated high benefit from MBS seen in clinics with the BMI-CDS intervention will be more likely than patients seen in usual care clinics to receive a referral to MBS
Number of new prescriptions of an FDA-approved pharmaceutical for obesity management | Within 18 months of index visit date
  Patients seen in clinics with the BMI-CDS intervention will be more likely than patients seen in usual care clinics to receive to receive a new prescription medication for obesity management
Change in weight trajectory during 18-month post-intervention follow-up period | 18 months following the index visit
  The within-patient slope of weight measurements over the 18 months following the index visit will be less positive for those seen in BMI-CDS intervention versus usual care clinics.

SECONDARY OUTCOMES:
Likelihood of patient conversation with their pcc about weight loss | 6 months following index visit
  Relative to patients with an index clinical encounter at usual care clinics, those with an index clinical encounter at BMI-CDS clinics will be more likely have had a conversation with their PCC about weight loss.
Intentions to engage in weight loss | 6 months following index visit
  Relative to patients with an index visit at usual care clinics, those with an index clinical encounter at BMI-CDS clinics will report stronger intentions to engage in weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, MD MPH MA, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Medical Group, Minneapolis, Minnesota, United States